CLINICAL TRIAL: NCT02339454
Title: Efficacy of Extracorporeal Shockwave Myocardial Revascularization Therapy in Patients With Stable Angina Pectoris - A Randomized, Double Blind, Placebo Controlled, Multicenter Study
Brief Title: Efficacy of Extracorporeal Shockwave Myocardial Revascularization Therapy in Patients With Stable Angina Pectoris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evgeny Shkolnik, MD (Other)
Collaborators: Vilnius University (Other); Medispec (Industry)
Responsible Party: Sponsor-Investigator, Evgeny Shkolnik, MD, Professor, department of functional methods in internal medicine, Moscow State University of Medicine and Dentistry
Organization: Moscow State University of Medicine and Dentistry (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESMR-RCT-UP
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Stable Angina Pectoris
Keywords: Cardiac Shock wave therapy; stable angina; exercise tolerance
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment group (Active Comparator): Patients in this group receive actual shockwave therapy. Study treatment consists of 9 sessions, with 3 sessions per week 1, 5 and 9. 100 shocks are delivered per spot, 1200 shocks per session.
  During 1st treatment week ESMR will be delivered 3 times (every other day) to basal segments (2 spots in each wall in apical 4-, 2-, 3- chamber positions).
  During 2nd treatment week ESMR will be delivered 3 times (every other day) to middle segments (2 spots in each wall in apical 4-, 2-, 3- chamber positions).
  During 3rd treatment week ESMR will be delivered 3 times (every other day) to apical segments (2 spots in each wall in apical 4-, 2-, 3- chamber positions).
  Interventions: Device: Active treatment group
- Placebo group (Placebo Comparator): This group of patients undergoes the same procedure as the treatment group; however shockwaves are not delivered to the heart.
  Interventions: Device: Placebo group

INTERVENTIONS:
Device: Active treatment group — Energy Density - 0.09 mJ/mm2 Device: Active Applicator
  Other Names: Cardiospec; Extracorporeal Shockwave Myocardial Revascularization (ESMR); Extracorporeal Cardiac Shock wave therapy (CSWT)
  Arms: Active treatment group
Device: Placebo group — Placebo Applicator
  Arms: Placebo group

SUMMARY:
Low intensity shockwaves have been proven in animal and pilot clinical studies to induce local growth of new blood vessels. Small single-center clinical trials with shockwave therapy showed promising results in reducing angina symptoms, improving perfusion and contractility in patients with refractory angina and stress-induced ischemia on imaging test.

The hypothesis of this study is that shockwave therapy could improve angina symptoms and exercise tolerance in broader population of patients with stable angina regardless of imaging test results Study aims to demonstrate anti-anginal efficacy of Extracorporeal Shockwave Myocardial Revascularization Therapy (ESMR), on top of stable optimal medical treatment in patients with stable angina.

DETAILED DESCRIPTION:
Low intensity shockwaves (0.09 millijoule/mm2) are delivered to myocardial tissue. Shockwaves are created by a special generator and are focused using a shockwave applicator device. The treatment is guided by standard echocardiography equipment. The shockwaves are delivered in synchronization with Patient R-wave (ECG) to avoid arrhythmias. The treatment is painless.

At first, the patient undergoes modified Bruce treadmill test, to assess exercise induced ischemia.

Exercise induced ECG ischemia is defined as the new development of horizontal or down - sloping ST segment depression (≥1 mm at 60 ms after J point) versus baseline tracing.

Study treatment consists of 9 sessions, with 3 sessions per week 1, 5 and 9. 100 shocks are delivered per spot, 1200 shocks per session.

During 1st treatment week ESMR will be delivered 3 times (every other day) to basal segments (2 spots in each wall in apical 4-, 2-, 3- chamber positions).

During 2nd treatment week ESMR will be delivered 3 times (every other day) to middle segments (2 spots in each wall in apical 4-, 2-, 3- chamber positions).

During 3rd treatment week ESMR will be delivered 3 times (every other day) to apical segments (2 spots in each wall in apical 4-, 2-, 3- chamber positions).

The spots are localized by the ultra-sound device and the shockwaves are focused to this area. Several treatments are required for optimal results.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients (females of childbearing potential must be using adequate contraceptive precautions such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence or vasectomized partner).
* Patients aged ≥ 18 years.
* Patients with coronary artery disease confirmed by angiography, prior MI, prior revascularization (PCI, CABG) and with exercise angina not controlled by the optimal medical therapy.
* Patient should be on a stable dosage of medication used to treat angina for at least 4 weeks prior to enrollment.
* ST-segment depression ≥ 1mm during exercise ECG.
* Able and willing to sign informed consent and to comply with study procedures.
* Written informed consent prior to enrolment into the study.

Exclusion Criteria:

* Angina at rest.
* ECG abnormalities at rest (left bundle-branch block, resting ST-segment depression ≥ 1mm, digoxin therapy, WPW-syndrome).
* Planned coronary intervention or CABG within 6 months.
* Heart failure (class III or IV NYHA).
* Moderate-severe hypertension (SBP>160 mmHg and/or DBP>100 mmHg).
* Hypotension (SBP<100 mmHg).
* Acute coronary syndrome or coronary revascularization procedure within the prior 3 months before enrolment.
* Females who are pregnant or nursing.
* Any clinically relevant hematological or biochemical abnormality on routine screening, according to Investigator's judgment.
* Severe concurrent pathology, including terminal illness (cancer, AIDS, etc.).
* Renal impairment defined as Creatinine >150 mcmol/l.
* Mild, moderate or severe hepatic impairment or hepatic insufficiency defined as: SGOT or SGPT > 3 times greater than normal upper limit or total serum bilirubin > 1.5 times greater than normal upper limit
* Existing contraindications for exercise testing (e.g. acute myocarditis or pericarditis, DVT, severe aortic stenosis)
* Dementia, psychosis, alcoholism (>350 g ethanol/week) or chronic abuse of medicines, drugs or psychoactive substances.
* Conditions which in the Investigator's opinion may interfere with the study's execution or due to which the patient should not participate for safety reasons.
* Risk of low patient cooperation.
* Inability or unwillingness to issue the informed consent.
* Patient is simultaneously participating in another device or drug study, or has participated in any clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization, or any cardiac shock wave therapy machine of a competitor company within 3 months of entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Exercise duration | 6 months
  To evaluate if ESMR able to improve total exercise duration in modified Bruce treadmill test.
  Patients will be assessed at baseline visit (screening) and 6 months after the first treatment.

SECONDARY OUTCOMES:
Time to 1 mm ST-segment depression in modified Bruce treadmill test | 6 months
Time to angina in modified Bruce treadmill test | 6 months
Number of angina attacks per week | 6 months
Number of sublingual nitroglycerin consumption per week | 6 months
CCS angina functional class | 6 months
Seattle angina questionnaire score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Celutkiene, MD, PhD, Principal Investigator — Vilnius University Hospital, Santariskiu klinikos; Evgeny Shkolnik, MD, PhD, Principal Investigator — Moscow State University of Medicine&Dentistry
Locations (2):
- Vilnius University Hospital, Santariskiu klinkos, Vilnius, Lithuania
- Moscow state university of medicine&dentistry, Moscow, Russia

REFERENCES:
- [Derived] Celutkiene J, Burneikaite G, Shkolnik E, Jakutis G, Vajauskas D, Cerlinskaite K, Zuoziene G, Petrauskiene B, Puronaite R, Komiagiene R, Butkuviene I, Steponeniene R, Misiura J, Laucevicius A. The effect of cardiac shock wave therapy on myocardial function and perfusion in the randomized, triple-blind, sham-procedure controlled study. Cardiovasc Ultrasound. 2019 Jul 4;17(1):13. doi: 10.1186/s12947-019-0163-1. PMID 31272465